CLINICAL TRIAL: NCT03087084
Title: RESpiration deTection From Implanted Cardiac Devices in Subjects With Heart Failure (REST-HF)
Acronym: REST-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: REST-HF
Record Dates: First submitted 2017-02-17; First posted 2017-03-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Pacing and Impedance Measurement system (Experimental)
  Interventions: Device: Cardiac Pacing and Impedance Measurement system

INTERVENTIONS:
Device: Cardiac Pacing and Impedance Measurement system — Subjects indicated for Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy Defibrillator device implant will be requested to perform some respiratory manoeuvres while impedance and electrogram signals are recorded by the system

SUMMARY:
The purpose of this prospective, non-randomized, single-arm, research study is to evaluate the accuracy of acutely extracting respiratory rate and tidal volume from implanted cardiac device impedance in subjects with heart failure.

In addition, to assess the feasibility of extracting respiratory rate from device EGM under various conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have heart failure and be undergoing implant of a new or replacement/upgrade Medtronic dual-chamber Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy Defibrillator device for approved indications;
* Subject must be implanted with an right ventricle lead that supports bipolar pacing and sensing (i.e. a true bipolar defibrillation lead);
* Subject must receive a light conscious sedation or no sedation where breathing maneuvers can be performed and evaluated during the implant;
* Subject must be willing to provide Informed Consent for their participation in the study;
* Subject must be ≥ 18 years of age.

Exclusion Criteria:

* Subjects who are unable or unwilling to voluntarily participate in any visit required by the study and to provide consent;
* Subject has congenital heart disease;
* Subject has a tachyarrhythmia (atrial and/or ventricular) at the time of enrollment and a cardioversion will not be attempted prior to the research procedure;
* Subject has unstable coronary artery disease;
* Subject requires cardiac pacing at rest for rate support;
* Subject presents any concomitant conditions which in the opinion of the investigator would not allow a proper execution of the respiratory exercises as per protocol;
* Subject presents any concomitant condition which in the opinion of the investigator would not allow a safe participation in the study;
* Subject is pregnant or breast feeding;
* Subject is legally incompetent;
* Subject is enrolled in a concurrent study that may confound the results of this study without documented pre-approval from Medtronic study manager.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of extracting respiratory features from intrathoracic impedance acutely in subjects with heart failure | Implant
  Impedance-derived respiratory rate during different breathing patterns

SECONDARY OUTCOMES:
Assess the feasibility of extracting respiratory rate from EGM under various conditions | Implant and 2 months follow-up
  EGM derived respiratory rate under various conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Van Heuverswyn, MD, Principal Investigator — University Ghent; Ashley Chin, MD, Principal Investigator — Groote Schuur Hospital; Hielko Miljoen, MD, Principal Investigator — University Hospital, Antwerp
Locations (3):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
- Groote Schuur Hospital, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No